CLINICAL TRIAL: NCT03414372
Title: Tough Talks: A Disclosure Intervention for HIV+ Young Men Who Have Sex With Men
Brief Title: Tough Talks: A Disclosure Intervention for HIV+ Young Men Who Have Sex With Men (YMSM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Virtually Better, Inc. (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-0345; 2R44MH104102-03 (NIH)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Hiv; HIV/AIDS; Disclosure
Keywords: MSM; HIV; disclosure; eHealth; virtual reality
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study includes 3 phases: 1) formative research to refine and enhance Tough Talks with input from YMSM and their social/sexual networks; 2) (n=8) a technical pilot to optimize functionality and technical performance; and 3) (n=156) a three-arm RCT to evaluate efficacy and effectiveness of Tough Talks among HIV-infected YMSM.
  In the RCT, the investigators will conduct a combined efficacy/effectiveness trial to compare the intervention delivered online, in the clinic or standard of care clinic messaging. Primary outcomes will be assessed at intervention completion (1 month) and at 6 months and include HIV viral load and condomless anal intercourse (CAI).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tough Talks Online (Experimental): Participants will use Tough Talks Online
  Interventions: Behavioral: Tough Talks Online
- Tough Talks Clinic (Experimental): Participants will use receive Tough Talks in a clinic
  Interventions: Behavioral: Tough Talks Clinic
- Standard of Care (Placebo Comparator): Participants will receive the standard of care (SOC).
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Tough Talks Online — Those randomized to the online condition will receive information about how to access Tough Talks online and be given their unique log-in and password information and information on how to contact study personnel for any technical issues. Arm 1 participants will have 24-hour access to all of the intervention features and will be able to access the program for additional sessions at any time. Study staff will provide reminders using text or email (participant preference) if they have not accessed the intervention at the specified time intervals.
  Other Names: Tough Talks
  Arms: Tough Talks Online
Behavioral: Tough Talks Clinic — Those randomized to the in-clinic condition (Arm 2) will immediately begin the Tough Talks intervention. Study staff will ensure participants are logged on and will also be available to answer technical issues should they arise. After completion, those in this arm will have an in-person follow-up visit scheduled for approximately two weeks. The in-person sessions were adapted to be delivered via Zoom or a similar HIPAA compliant platform due to the COVID-19 pandemic.
  Arms: Tough Talks Clinic
Behavioral: Standard of Care — Those randomized to the control arm (SOC) will receive a paper-based disclosure informational packet based on available Centers of Disease Control (CDC) guidance. At one-month, all participants will complete an online survey to assess intervention acceptability as well as to assess Social Cognitive Theory (SCT model) constructs.
  Arms: Standard of Care

SUMMARY:
Tough Talks is a virtual reality based HIV disclosure intervention that allows HIV+ individuals to practice disclosing to romantic partners. Tough Talks allows participants to have the opportunity to practice disclosing using a variety of strategies and experience different outcomes including acceptance, confusion, lack of HIV knowledge, and rejection.

DETAILED DESCRIPTION:
During Phase I of this project, the investigators developed an iPad based virtual reality system that features three avatars, two virtual locations and three disclosure scenarios which represent a variety of common disclosure experiences and contexts experienced by YMSM. In Phase II the investigators will further enhance Tough Talks and develop a full-feature automated version to test via a multi-site, randomized controlled trial (RCT) through the newly created Center for Innovative Technologies (iTech) across the Prevention and Care Continuum, an NIH-funded center to support adolescent HIV research.

ELIGIBILITY:
Inclusion Criteria:

* 16-29 years
* assigned male at birth
* male identified
* HIV infected
* Owns a mobile device or has access to a laptop or desktop computer
* able to understand, read, and speak English
* Reports 1 or more episodes of anal intercourse with a male partner in the last 6 months

Exclusion Criteria:

* HIV negative
* assigned female at birth
* 15 or younger
* 30 or older

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — assigned male sex at birth and currently male identified
Enrollment: 156 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Muessig, PhD, Principal Investigator — UNC-Chapel Hill; Lisa Hightow-Weidman, MD, Principal Investigator — UNC-Chapel Hll
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The investigators are not planning on making individual participant data available to other researchers.

REFERENCES:
- [Derived] Hightow-Weidman LB, Muessig K, Soberano Z, Rosso MT, Currie A, Adams Larsen M, Knudtson K, Vecchio A. Tough Talks Virtual Simulation HIV Disclosure Intervention for Young Men Who Have Sex With Men: Development and Usability Testing. JMIR Form Res. 2022 Sep 8;6(9):e38354. doi: 10.2196/38354. PMID 36074551

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Started | 53 | 51 | 52
Completed | 43 | 42 | 44
Not Completed | 10 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care | Total
Number analyzed (Participants) | 53 | 51 | 52 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.19 (3.50) | 23.92 (3.35) | 24.23 (3.46) | 23.78 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 53 | 51 | 52 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 13 | 41
  Not Hispanic or Latino | 38 | 38 | 39 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 32 | 33 | 28 | 93
  White | 13 | 11 | 13 | 37
  More than one race | 4 | 1 | 10 | 15
  Unknown or Not Reported | 2 | 3 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 51 | 52 | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suppressed Viral Load
Description: Chart review or drawn for study. Viral load suppression will be defined as HIV RNA < lower limit of detection as per the laboratory at each clinical site.
Time Frame: Month 6
Population: Data are reported for those participants who had a Month 6 viral load assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 39 | 39 | 41
Participants | 29 | 31 | 30

2. Secondary Outcome: Number of Participants Who Had Condomless Anal Intercourse With a Potentially Susceptible Partner
Description: Number of participants at month 6 with >/= 1 act of condomless anal intercourse with a partner who is not known to be HIV-positive within the last 3 months.
Time Frame: Month 6
Population: Data are reported for those participants who completed Month 6 survey and for which non-missing data are present.
Measure: Count of Participants; unit: Participants
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 29 | 22 | 25
Participants | 11 | 6 | 8

3. Secondary Outcome: Mean Intention to Disclose Score
Description: Measured using the Intention to Disclose scale which asks a single item: "I plan on telling my HIV status to all of my new partners before we have sex" and is rated using a 5-point Likert-type response scale. Scores range from 1 to 5 where '1' is "Strongly agree" and '5' is "Strongly disagree. "Lower scores indicate increased intention to disclose.
Time Frame: Month 6
Population: Participants were free to choose not to answer this question. Data reported for all non-missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 40 | 40 | 40
score on a scale | 1.45 (0.50) | 1.33 (0.47) | 1.15 (0.36)

4. Secondary Outcome: Mean Disclosure Self-Efficacy Score
Description: Measure of perceived ability to disclose HIV-seropositive status to casual sex partners in six scenarios. Scores were summed with higher scores indicating increased perceived ability to disclose. Six Questions were asked using a 5 point Likert Scale: 1=Absolutely sure I cannot; 2=Somewhat sure I cannot; 3=Not sure; 4=Somewhat sure I can; and 5=Absolutely sure I can. Scores range from 6-30.
Time Frame: Month 6
Population: Participants could choose not to respond to any of the six questions. Responses for participants who chose not to respond to any of the six questions were not counted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 38 | 37 | 36
score on a scale | 22.89 (7.69) | 23.03 (6.54) | 25.64 (7.24)

5. Secondary Outcome: Mean Consequences of Disclosure (Cost) Score
Description: Measure of a participant's perceived negative consequences of disclosing of their HIV status to a partner (e.g., "Relationship would get bad", "Person would not want to be around me"), with higher scores indicating higher perceived negative consequences of disclosure. Eight Questions rated using a 4-point Likert Scale 1=Strongly disagree 2=Disagree 3=Agree 4=Strongly Agree. Scores range from 8 to 32.
Time Frame: Month 6
Population: Participants could choose not to respond to any of the eight questions. Responses for participants who chose not to respond to any of the eight questions were not counted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 43 | 42 | 40
score on a scale | 23.40 (8.19) | 24.07 (8.84) | 19.20 (8.95)

6. Secondary Outcome: Mean Consequences of Disclosure (Rewards) Score
Description: Measure of a participant's perceived positive consequences of disclosing of their HIV status to a partner (e.g., "Keep them safe from HIV", "Improve the relationship"), with higher scores indicating higher perceived positive consequences of disclosure. Ten Questions rated using a 4-point Likert Scale 1=Strongly disagree; 2=Disagree; 3=Agree; and 4=Strongly Agree. Scores range from 10-40.
Time Frame: Month 6
Population: Participants could choose not to respond to any of the ten questions. Responses for participants who chose not to respond to any of the ten questions were not counted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 36 | 34 | 32
score on a scale | 32.22 (6.02) | 34.18 (6.15) | 34.31 (5.35)

7. Secondary Outcome: Mean Disclosure Self-Regulation (Family) Score
Description: Measured using a single question: "How many of your immediate family members are not aware of your HIV status but to whom you want to disclose?" and rated using a 5-point Likert Scale: 1=None; 2=Some, but less than half; 3=About half; 4=More than half; and 5=All. Scores range from 1 to 5 with lower scores indicating increased disclosure behaviors.
Time Frame: Month 6
Population: Participants were free to choose not to answer this question. Data reported for all non-missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 42 | 37 | 34
score on a scale | 2.57 (1.53) | 2.51 (1.48) | 2.59 (1.58)

8. Secondary Outcome: Mean Disclosure Self-Regulation (Peers) Score
Description: Measured using a single question: "How many of your peers are not aware of your HIV status but to whom you want to disclose?" and rated using a 5-point Likert Scale: 1=None; 2=Some, but less than half; 3=About half; 4=More than half; and 5=All. Scores range from 1 to 5 with lower scores indicating increased disclosure behaviors.
Time Frame: Month 6
Population: Participants were free to choose not to answer this question. Data reported for all non-missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 41 | 39 | 36
score on a scale | 2.49 (1.49) | 2.33 (1.18) | 2.67 (1.49)

9. Secondary Outcome: Mean Disclosure Self-Regulation (Sexual Partners) Score
Description: Measured using a single question: "How many of your current and past sexual partners are not aware of your HIV status but to whom you want to disclose?" and rated using a 5-point Likert Scale: 1=None; 2=Some, but less than half; 3=About half; 4=More than half; and 5=All. Scores range from 1 to 5 with lower scores indicating increased disclosure behaviors.
Time Frame: Month 6
Population: Participants were free to choose not to answer this question. Data reported for all non-missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 39 | 37 | 34
score on a scale | 2.08 (1.40) | 1.68 (1.03) | 1.71 (1.22)

10. Secondary Outcome: Mean Disclosure Outcome Expectations (Self-Evaluative) Score
Description: Measure of how a participant anticipates their behavior impacts their feelings or assessment of HIV protective behaviors. Higher scores indicate a more favorable/stronger evaluation/endorsement of HIV protective behaviors. Participant's self-evaluation based on six questions using a 5-point Likert scale (1, strongly disagree to 5, strongly agree) ranging from 5 to 30.
Time Frame: Month 6
Population: Although the protocol was not amended to remove this assessment, this scale was not used as study staff anticipated the questions included may be offensive to young participants.
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Mean Disclosure Outcome Expectations (Hedonistic) Score
Description: Measure of how a participant anticipates their behavior impacts their feelings or assessment of sexual pleasure or sensuality. Lower scores indicate a more favorable/stronger evaluation/endorsement of HIV protective behaviors. Participant's self-evaluation based on three questions using a 5-point Likert scale (1, strongly disagree to 5, strongly agree) ranging from 3 to 15.
Time Frame: Month 6
Population: as for outcome 10
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent through study completion, a total of up to 7 months.
Arm/Group | Tough Talks Online | Tough Talks Clinic | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51 | 1/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT03414372/Prot_SAP_000.pdf